CLINICAL TRIAL: NCT01816984
Title: A Biomarker Driven Pilot Study of the Pan-class I PI3K Inhibitor NVP-BKM120 in Combination With Cetuximab in Patients With Recurrent/Metastatic Head and Neck Cancer
Brief Title: PI3K Inhibitor BKM120 and Cetuximab in Treating Patients With Recurrent or Metastatic Head and Neck Cancer
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Chicago (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 12-1972; NCI-2013-00586 (Registry Identifier: CTRP (Clinical Trial Reporting Program))
Record Dates: First submitted 2013-03-20; First posted 2013-03-22 (Estimated); Results first posted 2020-10-27 (Actual); Last update posted 2021-10-05 (Actual); Status verified 2021-09

CONDITIONS: Metastatic Squamous Neck Cancer With Occult Primary Squamous Cell Carcinoma; Recurrent Metastatic Squamous Neck Cancer With Occult Primary; Recurrent Salivary Gland Cancer; Recurrent Squamous Cell Carcinoma of the Hypopharynx; Recurrent Squamous Cell Carcinoma of the Larynx; Recurrent Squamous Cell Carcinoma of the Lip and Oral Cavity; Recurrent Squamous Cell Carcinoma of the Nasopharynx; Recurrent Squamous Cell Carcinoma of the Oropharynx; Recurrent Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Recurrent Verrucous Carcinoma of the Larynx; Recurrent Verrucous Carcinoma of the Oral Cavity; Salivary Gland Squamous Cell Carcinoma; Stage IV Squamous Cell Carcinoma of the Hypopharynx; Stage IV Squamous Cell Carcinoma of the Nasopharynx; Stage IVA Salivary Gland Cancer; Stage IVA Squamous Cell Carcinoma of the Larynx; Stage IVA Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVA Squamous Cell Carcinoma of the Oropharynx; Stage IVA Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVA Verrucous Carcinoma of the Larynx; Stage IVA Verrucous Carcinoma of the Oral Cavity; Stage IVB Salivary Gland Cancer; Stage IVB Squamous Cell Carcinoma of the Larynx; Stage IVB Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVB Squamous Cell Carcinoma of the Oropharynx; Stage IVB Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVB Verrucous Carcinoma of the Larynx; Stage IVB Verrucous Carcinoma of the Oral Cavity; Stage IVC Salivary Gland Cancer; Stage IVC Squamous Cell Carcinoma of the Larynx; Stage IVC Squamous Cell Carcinoma of the Lip and Oral Cavity; Stage IVC Squamous Cell Carcinoma of the Oropharynx; Stage IVC Squamous Cell Carcinoma of the Paranasal Sinus and Nasal Cavity; Stage IVC Verrucous Carcinoma of the Larynx; Stage IVC Verrucous Carcinoma of the Oral Cavity; Tongue Cancer
MeSH Terms: conditions — Salivary Gland Neoplasms; Squamous Cell Carcinoma of Head and Neck; Tongue Neoplasms | interventions — NVP-BKM120; Cetuximab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Arm I (BKM120 PO and cetuximab 500 mg IV 14 days) (Experimental): Patients receive PI3K inhibitor BKM120 PO QD 100 mg/day on days -7 to 0. Patients complete 1 week washout. 3 patients receive BKM120 PO 80mg / day and cetuximab 500 mg IV /14 days and after dose escalation, 9 patients receive BKM120 PO 100mg / day and cetuximab 500 mg IV /14 days thereafter.
  All patients receive PI3K inhibitor BKM120 PO QD day on days 1-28 and cetuximab IV over 60-120 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  Interventions: Drug: PI3K inhibitor BKM120; Biological: cetuximab

INTERVENTIONS:
Drug: PI3K inhibitor BKM120 — Given PO
  Other Names: BKM120; PI3K_Inhibitor_BKM120
Biological: cetuximab — Given IV
  Other Names: C225; C225 monoclonal antibody; IMC-C225; MOAB C225; monoclonal antibody C225

SUMMARY:
This pilot randomized phase I/II trial studies the side effects and best dose of PI3K inhibitor BKM120 when given together with cetuximab and to see how well it works in treating patients with recurrent or metastatic head and neck cancer. PI3K inhibitor BKM120 may stop the growth of tumor cells by blocking some of the enzymes needed for cell growth. Monoclonal antibodies, such as cetuximab, can block tumor growth in different ways. Some block the ability of tumors to grow and spread. Others find tumor cells and help kill them or carry tumor-killing substances to them. Giving PI3K inhibitor BKM120 together with cetuximab may kill more tumor cells

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Induction of compensatory signaling/feedback loop signaling after one week of BKM120 (PI3K inhibitor BKM120) (run-in) compared to patients not treated with BKM120.

II. Safety and tolerability of combined treatment with BKM120 and cetuximab.

SECONDARY OBJECTIVES:

I. Induction of apoptosis after one week of BKM120 (run-in) compared to patients not treated with BKM.

II. Tumor shrinkage (based Response Evaluation Criteria in Solid Tumors [RECIST] version 1.1 [V1.1] measurements) in patients treated with combination.

III. Response rate (based RECIST V1.1 measurements) in patients treated with combination.

IV. Overall survival. V. Progression free survival.

OUTLINE: This is a phase I, dose-escalation study of PI3K inhibitor BKM120, followed by a phase II study.

RUN-IN-PERIOD: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive PI3K inhibitor BKM120 orally (PO) once daily (QD) on days -7 to 0. Patients complete 1 week washout before dose escalation.

ARM II: Patients receive no treatment on days -7 to 0.

All patients receive PI3K inhibitor BKM120 PO QD on days 1-28 and cetuximab intravenously (IV) over 60-120 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up for 28 days.

ELIGIBILITY:
Inclusion Criteria:

* Histologically / cytologically confirmed diagnosis of squamous cell carcinoma of head and neck origin not amenable to curative intent therapy; both human papillomavirus (HPV)(+) and HPV(-) tumors are eligible; tumors (squamous histology) of unknown primary that are clearly related to the head and neck area are eligible
* Presence of measurable lesions (RECIST V1.1)
* Mandatory tumor biopsy/biopsies in accessible tumors; for inaccessible tumors availability of tissue is required: >= 10 tumor containing formalin-fixed paraffin-embedded (FFPE) slides/sections
* Progressive disease after exposure to a platinating agent (e.g. cisplatin or carboplatin) in a prior line of therapy, or documented intolerance to such an agent
* Eastern Cooperative Oncology Group (ECOG) performance status =< 2
* No more than two lines of prior cytotoxic chemotherapy in the recurrent/metastatic (palliative intent) treatment setting
* Prior use of cetuximab or another epidermal growth factor receptor (EGFR) inhibitor is allowable and if used as a single agent should not be considered as a cytotoxic chemotherapy
* Patients must have at least one site of measurable disease (if applicable) (per RECIST for solid tumors or the appropriate disease classification/criteria for the target population)
* Absolute neutrophil count (ANC) >= 1.5 x 10^9/L
* Platelets >= 100 x 10^9/L
* Hemoglobin (Hb) > 9 g/dL
* Total calcium (corrected for serum albumin) within normal limits
* Magnesium >= the lower limit of normal for the institution
* Potassium within normal limits for the institution
* Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) within 1.5 x normal range (or =< 3.0 x upper limit of normal [ULN] if liver metastases are present)
* Serum bilirubin within normal range (or =< 1.5 x ULN if liver metastases are present; or total bilirubin =< 3.0 x ULN with direct bilirubin within normal range in patients with well documented Gilbert syndrome)
* Serum creatinine =< 1.5 x ULN or 24-hour clearance >= 50 mL/min
* Serum amylase =< ULN
* Serum lipase =< ULN
* Fasting plasma glucose =< 120 mg/dL (6.7 mmol/L)
* Negative serum pregnancy test within 72 hours before starting study treatment in women with childbearing potential
* Signed informed consent
* International normalized ratio (INR) =< 2.5

Exclusion Criteria:

* Patients who have received prior treatment with a P13K inhibitor
* No available tumor material for correlative studies
* Patients with a known hypersensitivity to BKM120 or to its excipients, or hypersensitivity to cetuximab
* More than two prior lines of cytotoxic chemotherapy in the recurrent/metastatic disease setting (palliative treatment intent)(excluding single agent use of an EGFR inhibitor)
* Patients with untreated brain metastases are excluded; however, patients with treated brain metastases are eligible if they are > 4 weeks from therapy completion (including radiation and/or surgery), are clinically stable at the time of study entry and are not receiving corticosteroid therapy at the time of study entry
* Patients with acute or chronic liver, renal disease or pancreatitis
* Patients with the following mood disorders as judged by the Investigator or a psychiatrist, or as a result of patient's mood assessment questionnaire (treating physician to decide on whether to administer questionnaire):

  * Medically documented history of or active major depressive episode, bipolar disorder (I or II), obsessive-compulsive disorder, schizophrenia, a history of suicidal attempt or ideation, or homicidal ideation (immediate risk of doing harm to others)
  * >= Common Terminology Criteria for Adverse Events (CTCAE) version 4 (v4) grade 3 anxiety
  * Meets the cut-off score of >= 10 in the Patient Health Questionnaire 9 (PHQ-9) or a cut-off of >= 15 in the Generalized Anxiety Disorder 7 (GAD-7) mood scale, respectively, or selects a positive response of "1, 2, or 3" to question number 9 regarding potential for suicidal thoughts in the PHQ-9 (independent of the total score of the PHQ-9)
* Patients with diarrhea >= CTCAE v4 grade 2
* Patient has active cardiac disease including any of the following:

  * History of clinically significant heart failure (previously assessed) with a left ventricular ejection fraction (LVEF) of < 50% as determined by multiple grated acquisition (MUGA) scan or echocardiogram (ECHO)
  * Corrected QT (QTc) > 480 msec on screening electrocardiogram (ECG) (using the Fridericia QT correction [QTcF] formula)
  * Angina pectoris that requires the use of anti-anginal medication
  * Ventricular arrhythmias except for benign premature ventricular contractions
  * Supraventricular and nodal arrhythmias requiring a pacemaker or not controlled with medication
  * Conduction abnormality requiring a pacemaker
  * Valvular disease with document compromise in cardiac function
  * Symptomatic pericarditis
* Patient has a history of cardiac dysfunction including any of the following:

  * Myocardial infraction within the last 6 months, documented by persistent elevated cardiac enzymes or persistent regional wall abnormalities on assessment of LVEF function
  * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
  * Documented cardiomyopathy
* Patient has poorly controlled diabetes mellitus or steroid-induced diabetes mellitus (hemoglobin A1C [HbA1C] > 7.5%)
* Patients with any history of hyperglycemia (elevated blood glucose level on blood chemistries) should be considered for initiation of Metformin treatment (500mg, PO, twice daily) prior to starting BKM120
* Other concurrent severe and/or uncontrolled concomitant medical conditions (e.g., active or uncontrolled infection) that could cause unacceptable safety risks or compromise compliance with the protocol

  * Significant symptomatic deterioration of lung function; if clinically indicated, pulmonary function tests including measures of predicted lung volumes, diffusing capacity of the lung for carbon monoxide (DLCO), oxygen (O2) saturation at rest on room air should be considered to exclude pneumonitis or pulmonary infiltrates
* Impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of BKM120 (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection); patients with unresolved diarrhea will be excluded as previously indicated
* Patients who have been treated with any hematopoietic colony-stimulating growth factors (e.g., filgrastim [G-CSF], sargramostim [GM-CSF]) =< 2 weeks prior to starting study drug; erythropoietin or darbepoetin therapy, if initiated at least 2 weeks prior to enrollment, may be continued
* Patients who are currently receiving treatment with medication with a known risk to prolong the QT interval or inducing Torsades de Pointes and the treatment cannot either be discontinued or switched to a different medication prior to starting study drug
* Patients receiving chronic treatment with steroids or another immunosuppressive agent other than specified in exclusion criterion #4

  * Note: Topical applications (e.g. rash), inhaled sprays (e.g. obstructive airways diseases), eye drops or local injections (e.g. intra-articular) are allowed; patients with previously treated brain metastases, who are on stable low dose corticosteroids treatment (eg. dexamethasone 2 mg/day, prednisolone 10 mg/day) for at least 14 days before start of study treatment are eligible
* Patients who have taken herbal medications and certain fruits within 7 days prior to starting study drug; herbal medications include, but are not limited to St. John's wort, Kava, ephedra (ma huang), gingko biloba, dehydroepiandrosterone (DHEA), yohimbe, saw palmetto, and ginseng; fruits include the cytochrome P450, family 3, subfamily A (CYP3A) inhibitors Seville oranges, grapefruit, pummelos, or exotic citrus fruits
* Patients who are currently treated with drugs known to be moderate and strong inhibitors or inducers of isoenzyme CYP3A, and the treatment cannot be discontinued or switched to a different medication prior to starting study drug
* Patients who have received chemotherapy or targeted anticancer therapy =< 4 weeks (6 weeks for nitrosourea, antibodies or mitomycin-C) prior to starting study drug must recover to a grade 1 before starting the trial
* Patients who have received any continuous or intermittent small molecule therapeutics (excluding monoclonal antibodies) =< 5 effective half lives prior to starting study drug or who have not recovered from side effects of such therapy; typically a >= 2 week interval since completion of prior therapy is recommended and 4 weeks for monoclonal antibodies
* Patients who have received wide field radiotherapy =< 4 weeks or limited field radiation for palliation =< 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who have undergone major surgery =< 2 weeks prior to starting study drug or who have not recovered from side effects of such therapy
* Patients who are currently taking therapeutic doses of warfarin sodium or any other Coumadin-derivative anticoagulant
* Women who are pregnant or breast-feeding or adults of reproductive potential not employing an effective method of birth control; double barrier contraceptives must be used through the trial by both sexes; oral, implantable, or injectable contraceptives may be affected by cytochrome P450 interactions, and are therefore not considered effective for this study; women of child-bearing potential, defined as sexually mature women who have not undergone a hysterectomy or who have not been naturally postmenopausal for at least 12 consecutive months (i.e., who has had menses any time in the preceding 12 consecutive months), must have a negative serum pregnancy test =< 72 hours prior to initiating treatment
* Known diagnosis of human immunodeficiency virus (HIV) infection unless patient is fully immunocompetent (cluster of differentiation 4 [CD4] > 200) and patient is not taking antiretroviral therapy
* History of another malignancy within 3 years, except cured basal cell carcinoma of the skin or excised carcinoma in situ of the cervix, or any tumor that is after clearing with the principal investigator (PI) clearly not considered to have impact on prognosis
* Patient is unable or unwilling to abide by the study protocol or cooperate fully with the investigator

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2013-05; Primary Completion 2018-04 (Actual); Study Completion 2020-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Tanguy Seiwert, Principal Investigator — University of Chicago Comprehensive Cancer Center
Locations (1):
- University of Chicago Comprehensive Cancer Center, Chicago, Illinois, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Arm I (BKM120 PO and Cetuximab 500 mg IV 14 Days): Patients receive PI3K inhibitor BKM120 PO QD 100 mg/day on days -7 to 0. Patients complete 1 week washout. After dose escalation phase, 3 patients receive BKM120 PO 80mg / day and cetuximab 500 mg IV /14 days and 9 patients receive BKM120 PO 100mg / day and cetuximab 500 mg IV /14 days thereafter.
  All patients receive PI3K inhibitor BKM120 PO QD day on days 1-28 and cetuximab IV over 60-120 minutes on days 1 and 15. Courses repeat every 28 days in the absence of disease progression or unacceptable toxicity.
  PI3K inhibitor BKM120: Given PO
  cetuximab: Given IV
Period: Overall Study
Arm/Group | Arm I (BKM120 PO and Cetuximab 500 mg IV 14 Days)
Started | 12
Completed | 11
Not Completed | 1
Not completed — declining health status | 1

BASELINE CHARACTERISTICS:
Arm/Group | Arm I (BKM120 PO and Cetuximab 500 mg IV 14 Days)
Number analyzed (Participants) | 12
Age, Continuous [Median (Full Range); unit: years] | 61 [47 to 73]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2
  Male | 10
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 11
  African American | 1
Region of Enrollment [Number; unit: participants]
  United States | 12

OUTCOME MEASURES:

1. Primary Outcome: Compensatory Signaling/Feedback Loop Signaling Evaluated by Measurement of Phosphorylated (p)-EGFR
Description: Performed using snap frozen tissue samples using the well-established PamGene Kinase array platform available in the Salgia/Seiwert laboratories.
Time Frame: 1 week
Population: Data not collected
Arm/Group | Arm I (BKM120 PO and Cetuximab 500 mg IV 14 Days)
Number analyzed (Participants) | 0

2. Primary Outcome: Maximum Tolerated Dose (MTD)
Description: Maximum tolerated dose (MTD) is defined as the dose level preceding the dose in which greater than or equal to 2 out of 3-6 patients experience a dose limiting toxicity (DLT) assessed using CTCAE v4
Time Frame: 28 days
Population: 0 patients out of 3 from the BKM 80mg/day cohort had DLT (dose limiting toxicities). 0 patients out of 9 from the BKM 100mg/day cohort had DLT.
Measure: Number; unit: mg / day
Arm/Group | Arm I (BKM120 PO and Cetuximab 500 mg IV 14 Days)
Number analyzed (Participants) | 12
mg / day | 100

3. Secondary Outcome: Apoptosis Induction
Description: Measured by Terminal deoxynucleotidyl transferase dUTP nick end labeling (TUNEL) assay on Formalin-Fixed, Paraffin-Embedded (FFPE) sections in a descriptive manner.
Time Frame: Up to 28 days
Population: Data not collected.
Arm/Group | Arm I (BKM120 PO and Cetuximab 500 mg IV 14 Days)
Number analyzed (Participants) | 0

4. Secondary Outcome: Response Rate Assessed Using RECIST
Description: Percentage of patients whose cancer shrinks or disappears after treatment.
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (BKM120 PO and Cetuximab 500 mg IV 14 Days)
Number analyzed (Participants) | 12
Participants | 1

5. Secondary Outcome: Response Rate in Patients With Prior EGFR Failure Assessed Using RECIST
Description: Percentage of patients with prior EGFR failure assessed using RECIST whose cancer shrinks or disappears after treatment.
Time Frame: Up to 28 days
Measure: Count of Participants; unit: Participants
Arm/Group | Arm I (BKM120 PO and Cetuximab 500 mg IV 14 Days)
Number analyzed (Participants) | 11
Participants | 1

6. Secondary Outcome: Tumor Shrinkage
Description: Tumor shrinkage will be visualized as a waterfall plot for graphical (qualitative) comparison.
Time Frame: Up to 28 days
Population: Data not collected.
Arm/Group | Arm I (BKM120 PO and Cetuximab 500 mg IV 14 Days)
Number analyzed (Participants) | 0

7. Secondary Outcome: Overall Survival
Description: Overall survival is defined as the time from study initiation to death due to any reason.
Time Frame: 4 years and 3 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (BKM120 PO and Cetuximab 500 mg IV 14 Days)
Number analyzed (Participants) | 12
months | 9.3 [5.5 to 14]

8. Secondary Outcome: Progression Free Survival
Description: Progression free survival is defined as the time from study initiation to first evidence of progression of disease.
Time Frame: 4 years and 3 months
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Arm I (BKM120 PO and Cetuximab 500 mg IV 14 Days)
Number analyzed (Participants) | 12
months | 2 [1.7 to 5]

ADVERSE EVENTS:
Time Frame: 4 years and 3 months
Arm/Group | Arm I (BKM120 PO and Cetuximab 500 mg IV 14 Days)
All-Cause Mortality (participants affected / at risk) | 12/12
Serious Adverse Events (participants affected / at risk) | 4/12
Other Adverse Events (participants affected / at risk) | 12/12
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (BKM120 PO and Cetuximab 500 mg IV 14 Days) (N=12)
Electrolyte abnormality and anemia (Metabolism and nutrition disorders) | 1
Orthostatis (Vascular disorders) | 1
Acute Kidney Injury (Renal and urinary disorders) | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (BKM120 PO and Cetuximab 500 mg IV 14 Days) (N=12)
Hyperglycemia (Metabolism and nutrition disorders) | 11
Hypomagnesemia (Metabolism and nutrition disorders) | 10
Anorexia (Gastrointestinal disorders) | 8
Fatigue (General disorders) | 8
Pain (General disorders) | 8
Hypoalbuminemia (Metabolism and nutrition disorders) | 7
Rash (Skin and subcutaneous tissue disorders) | 7
ALT Increase (Metabolism and nutrition disorders) | 7
AST increase (Metabolism and nutrition disorders) | 6
Diarrhea (Gastrointestinal disorders) | 6
Hypokalemia (Metabolism and nutrition disorders) | 5
Anxiety (Nervous system disorders) | 4
Constipation (Gastrointestinal disorders) | 4
Mood changes (General disorders) | 3
Mucositis (Gastrointestinal disorders) | 3
Nausea (Gastrointestinal disorders) | 3
Pruritis (Skin and subcutaneous tissue disorders) | 3
Transaminitis (General disorders) | 3
Anemia (General disorders) | 2
Dysphagia (Gastrointestinal disorders) | 2
Increased BUN (Metabolism and nutrition disorders) | 2
Leg tremor (General disorders) | 2
Total bilirubin increase (Blood and lymphatic system disorders) | 2
Vomiting (Gastrointestinal disorders) | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2014-02-16): https://cdn.clinicaltrials.gov/large-docs/84/NCT01816984/Prot_SAP_000.pdf